CLINICAL TRIAL: NCT04316208
Title: The Effect of Intraoperative Variations in Positive-End Expiratory Pressure on Subdural Pressure, Optic Nerve Sheath Diameter, Lung Compliance and Brain Perfusion Pressure in Supratentorial Tumor Surgery
Brief Title: Effect of PEEP on Subdural Pressure, Optic Nerve Sheath Diameter, Lung Compliance and Brain Perfusion Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Özlem Korkmaz Dilmen, Professor in Anesthesiology and Reanimation, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ST_18032020
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Supratentorial Neoplasms; Anesthesia, General; Optic Nerve
MeSH Terms: conditions — Supratentorial Neoplasms

STUDY DESIGN:
Intervention Model Description: After craniotomy, PEEP will be adjusted to 0 cmH2O, 5 cmH2O and 10 cmH2O for 5 minutes each to collect the data
Masking Description: Care provider will adjust the PEEP level, make measurements and record arterial blood gas analysis results. Biostatistician will compare data set at each PEEP to each other. Investigator will analyze the data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supratentorial tumor surgery (Experimental): Patients undergoing elective supratentorial tumor surgery under general anesthesia will be ventilated with positive end-expiratory pressures of 0, 5 and 10 cmH2O after craniotomy.
  Interventions: Procedure: PEEP variations

INTERVENTIONS:
Procedure: PEEP variations — Patients will be ventilated with a PEEP of 5 cmH2O during induction of anesthesia. After craniotomy, the PEEP will be reduced to 0 cmH2O for 5 minutes and data will be collected at the end of 5 minutes. Next, PEEP will be increased to 5 cmH2O for 5 minutes and data will be collected at the end of 5 minutes. Finally, PEEP will be increased to 10 cmH2O for 5 minutes and data will be collected at the end of 5 minutes.

SUMMARY:
We aim to determine the level of intraoperative PEEP that optimizes lung compliance without causing a rise in subdural pressure and if we can utilize optic nerve sheath diameter measurement as an indicator for ICP while optimizing lung compliance during supratentorial tumor surgeries.

DETAILED DESCRIPTION:
Application of positive end-expiratory pressure (PEEP) during general anesthesia minimizes ventilation/perfusion mismatch, intraoperative atelectasis and postoperative pulmonary complications. PEEP application in intracranial surgeries is usually avoided due to the risk of raised intracranial pressure (ICP) leading to decreased cerebral perfusion pressure (CPP). Several studies examine the effects of PEEP on subdural pressure and CPP however none examine how lung compliance is affected at the same time. Ultrasound-guided measurement of optic nerve sheath diameter (ONSD) is an indirect indicator of raised ICP and there is limited literature on the correlation of ONSD and ICP during intracranial surgery. In this study, we aim to determine the level of intraoperative PEEP that optimizes lung compliance without causing a rise in subdural pressure and if we can utilize ONSD measurement as an indicator for ICP while optimizing lung compliance during supratentorial tumor surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Supratentorial tumor
* Elective surgery
* American Society of Anesthesiologist Class I, II or III

Exclusion Criteria:

* Midline shift more than 5 mm determined by intracranial imaging
* Initial subdural pressure higher than 20 mmHg
* Requiring intravenous mannitol or hypertonic saline treatment before dural opening
* Congestive heart failure
* Pulmonary hypertension
* Sepsis
* Hypovolemia
* Obstructive or restrictive lung disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Subdural pressure | Measurements will look at the change between 3 timepoints: at 5 minutes with PEEP of 0 cmH2O (T0), then at 5 minutes with PEEP of 5 cmH2O (T5), and finally at 5 minutes with PEEP of 10 cmH2O (T10)
  22G/ 0.9mm catheter will be introduced into subdural space after craniotomy and connected to the transducer for pressure measurement
Optic nerve sheath diameter (left and right) | Measurements will look at the change between 3 timepoints: at 5 minutes with PEEP of 0 cmH2O (T0), then at 5 minutes with PEEP of 5 cmH2O (T5), and finally at 5 minutes with PEEP of 10 cmH2O (T10)
  Ultrasound-guided measurement with the linear probe.

SECONDARY OUTCOMES:
Mean arterial pressure | Measurements will look at the change between 3 timepoints: at 5 minutes with PEEP of 0 cmH2O (T0), then at 5 minutes with PEEP of 5 cmH2O (T5), and finally at 5 minutes with PEEP of 10 cmH2O (T10)
  Invasive blood pressure monitoring will be done. The transducer will be kept at the same level as the transducer for the subdural pressure, at the level of the external ear canal
Brain relaxation index | Measurements will look at the change between 3 timepoints: at 5 minutes with PEEP of 0 cmH2O (T0), then at 5 minutes with PEEP of 5 cmH2O (T5), and finally at 5 minutes with PEEP of 10 cmH2O (T10)
  1: dura is under the cranium, 2: dura is at the level of the cranium, 3: dura is above the cranium 4: dural pulsations ceased
Arterial blood gases | Measurements will look at the change between 3 timepoints: at 5 minutes with PEEP of 0 cmH2O (T0), then at 5 minutes with PEEP of 5 cmH2O (T5), and finally at 5 minutes with PEEP of 10 cmH2O (T10)
  Arterial oxygen pressure and arterial carbon dioxide pressure will be recorded
Regional cerebral oxygen saturation | Measurements will look at the change between 3 timepoints: at 5 minutes with PEEP of 0 cmH2O (T0), then at 5 minutes with PEEP of 5 cmH2O (T5), and finally at 5 minutes with PEEP of 10 cmH2O (T10)
  % - measurement taken with INVOS cerebral oximeter
Lung compliance | Measurements will look at the change between 3 timepoints: at 5 minutes with PEEP of 0 cmH2O (T0), then at 5 minutes with PEEP of 5 cmH2O (T5), and finally at 5 minutes with PEEP of 10 cmH2O (T10)
  L/cmH2O - measurement taken from Draeger Dräger Perseus® A500 mechanical ventilator

OTHER OUTCOMES:
P/F ratio | Measurements will look at the change between 3 timepoints: at 5 minutes with PEEP of 0 cmH2O (T0), then at 5 minutes with PEEP of 5 cmH2O (T5), and finally at 5 minutes with PEEP of 10 cmH2O (T10)
  Obtained by PaO2/FiO2. Hence FiO2 will be recorded at the times of measurements
Brain perfusion pressure | Measurements will look at the change between 3 timepoints: at 5 minutes with PEEP of 0 cmH2O (T0), then at 5 minutes with PEEP of 5 cmH2O (T5), and finally at 5 minutes with PEEP of 10 cmH2O (T10)
  Calculated from subdural pressure and mean arterial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Tunali, MD, Principal Investigator — Istanbul University Cerrahpasa Medical Faculty
Locations (1):
- Istanbul University - Cerrahpasa, Department of Neurosurgery, Neurosurgical Theaters, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Caricato A, Conti G, Della Corte F, Mancino A, Santilli F, Sandroni C, Proietti R, Antonelli M. Effects of PEEP on the intracranial system of patients with head injury and subarachnoid hemorrhage: the role of respiratory system compliance. J Trauma. 2005 Mar;58(3):571-6. doi: 10.1097/01.ta.0000152806.19198.db. PMID 15761353
- [Background] Mascia L, Grasso S, Fiore T, Bruno F, Berardino M, Ducati A. Cerebro-pulmonary interactions during the application of low levels of positive end-expiratory pressure. Intensive Care Med. 2005 Mar;31(3):373-9. doi: 10.1007/s00134-004-2491-2. Epub 2005 Jan 25. PMID 15668765
- [Background] Flexman AM, Gooderham PA, Griesdale DE, Argue R, Toyota B. Effects of an alveolar recruitment maneuver on subdural pressure, brain swelling, and mean arterial pressure in patients undergoing supratentorial tumour resection: a randomized crossover study. Can J Anaesth. 2017 Jun;64(6):626-633. doi: 10.1007/s12630-017-0863-7. Epub 2017 Mar 24. PMID 28342045
- [Background] Corradi F, Robba C, Tavazzi G, Via G. Combined lung and brain ultrasonography for an individualized "brain-protective ventilation strategy" in neurocritical care patients with challenging ventilation needs. Crit Ultrasound J. 2018 Sep 17;10(1):24. doi: 10.1186/s13089-018-0105-4. PMID 30221312
- [Background] Rasmussen M, Bundgaard H, Cold GE. Craniotomy for supratentorial brain tumors: risk factors for brain swelling after opening the dura mater. J Neurosurg. 2004 Oct;101(4):621-6. doi: 10.3171/jns.2004.101.4.0621. PMID 15481716
- [Background] Ruggieri F, Beretta L, Corno L, Testa V, Martino EA, Gemma M. Feasibility of Protective Ventilation During Elective Supratentorial Neurosurgery: A Randomized, Crossover, Clinical Trial. J Neurosurg Anesthesiol. 2018 Jul;30(3):246-250. doi: 10.1097/ANA.0000000000000442. PMID 28671879